CLINICAL TRIAL: NCT06764264
Title: Cognitive Assessment During Heat Tolerance Test
Brief Title: Integrating Cognitive Assessments Into the Heat Tolerance Test After Exertional Heat Injury
Status: Completed | Type: Observational
Sponsor: Medical Corps, Israel Defense Force (Other)
Collaborators: The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, ITAY, Dr. Sagi Shpitzer, MD, Chief Medical Officer, IDF Physiology Institute, Principal Investigator, Medical Corps, Israel Defense Force
Other Study IDs: IDF- 123 1779-2017
Record Dates: First submitted 2024-12-24; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Exertional Heat Injury
Keywords: Heat Tolerance Test; Exertional heat injury; Cognitive Impairment; Thermoregulatory Function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Combat soldiers post exertional heat injury: Participants were classified into heat-intolerant (HI) or heat-tolerant (HT) groups based on their HTT physiological outcomes.

SUMMARY:
This prospective observational study is to evaluate soldiers post-exertional heat injury (EHI) during a heat tolerant test (HTT) to investigate the impact on their cognitive performance.

DETAILED DESCRIPTION:
The objective of the proposed research is to add a cognitive evaluation to the physiological parameters monitored in the heat tolerance test (HTT) and to construct a new cognitive-physiological model for evaluation based on the accumulated knowledge on soldiers' heat tolerance. Each year, in the Israel Defense Forces (IDF), approximately 50 soldiers post exertional heat injury (EHI) are referred to perform the HTT. The HTT is carried out approximately one month post injury as part of clinical evaluation of the patient and is also intended to determine return to duty for combatants in field units. Currently, the criteria used in the HTT to determine heat tolerance are based solely on physiological parameters, while no cognitive evaluation is utilized in the HTT. Noteworthy are the numerous studies published in scientific literature describing the influence of exposure to heat conditions and physical effort on cognition and psychological strain in humans.

The subjects performing the HTT will also undergo cognitive evaluation and psychological strain assessment using tests used and validated in the research laboratories of the United States military (USARIEM). The cognitive evaluation will be performed in addition to the validated physiological monitoring performed in the HTT. All gathered physiological and cognitive data will be used to construct new bio-statistical models and new criteria will be suggested for the definition of heat tolerance or intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Combat soldiers post exertional heat injury

Exclusion Criteria:

* Additional medical condition restricting combat duty

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Israeli Defense Forces combat soldiers
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants Classified as Heat-Intolerant during Heat Tolerant Test | 120 minutes
  Participants are classified as heat-intolerant if they exhibit any of the following indicators during the Heat Tolerance Test: a core body temperature (Tre) ≥ 38.5°C (≥ 101.38°F), a heart rate (HR) ≥ 150 bpm, or failure to achieve a Tre-to-HR ratio ≥ 0.2798°C ∙ bpm-¹. Participants meeting none of these criteria are classified as heat-tolerant.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Moran, PhD, Study Director — Institute of Military Physiology, IDF Medical Corps, Tel Hashomer, Israel
Locations (1):
- Heller Institute, Institute of Military Physiology, IDF Medical Corps, Tel Litwinsky, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
The data for this belong to the Israel Defense Forces and the Israel Ministry of Defense. Data sharing will be considered if the corresponding author receives a reasonable request and establishes an institution-to-institution data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data are available, and sharing will be considered if the corresponding author receives a reasonable request and establishes an institution-to-institution data-sharing agreement.
Access Criteria: Sharing will be considered if the corresponding author receives a reasonable request and establishes an institution-to-institution data-sharing agreement.

REFERENCES:
- [Background] Moran DS, Shitzer A, Pandolf KB. A physiological strain index to evaluate heat stress. Am J Physiol. 1998 Jul;275(1):R129-34. doi: 10.1152/ajpregu.1998.275.1.R129. PMID 9688970
- [Background] Epstein Y, Sohar E, Shapiro Y. Exertional heatstroke: a preventable condition. Isr J Med Sci. 1995 Jul;31(7):454-62. PMID 7607879
- [Background] Moran DS, Heled Y, Still L, Laor A, Shapiro Y. Assessment of heat tolerance for post exertional heat stroke individuals. Med Sci Monit. 2004 Jun;10(6):CR252-7. Epub 2004 Jun 1. PMID 15173669
- [Background] Moran DS, Erlich T, Epstein Y. The heat tolerance test: an efficient screening tool for evaluating susceptibility to heat. J Sport Rehabil. 2007 Aug;16(3):215-21. doi: 10.1123/jsr.16.3.215. PMID 17923727